CLINICAL TRIAL: NCT06285292
Title: Prospective and Comparative Evaluation of a Medical Device Composed of a Perineal Probe Connected to a Mobile Application in the Management of Stress Urinary Incontinence.
Acronym: PRIME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: FIZIMED Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC24_0097
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence, pelvic-floor muscles, pelvic-perineal rehabilitation
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMY (connected biofeedback medical device) (Experimental): 2 rehabilitation between M0 and M2 and pelvic-perineal exercises with the EMY device on 3 different days a week, for 15 minutes, over a period of 3 months.
  Interventions: Device: EMY
- standard (No Intervention): 15 sessions of pelvic floor rehabilitation (gold standard)

INTERVENTIONS:
Device: EMY — Patients in the "intervention" group (rehabilitation with the EMY medical device) will undergo 2 rehabilitation sessions with a physiotherapist trained in pelviperineology between M0 and M2. The aim of these sessions will be to learn proper perineal contraction and combat the deficits identified during the physiotherapist's assessment. They will have to perform pelvic-perineal re-education exercises with the EMY device on 3 different days a week, for 15 minutes, over a period of 3 months. Then, for a further 3 months, their program can be modified for free, on-demand use (e.g. 2 x 10 minutes per week). After the main criterion at M6, they will be free to modify their rehabilitation program in the application according to their symptoms, and follow their program until the end of the study
  Other Names: pelvic-perineal probe
  Arms: EMY (connected biofeedback medical device)

SUMMARY:
Stress urinary incontinence (SUI) affects around 40% of women and has a major impact on quality of life. The gold standard for the treatment of SUI is pelvicfloor rehabilitation, but this presents constraints in terms of availability of healthcare professionals, as well as organization and travel for patients. Innovative devices offer self-training exercises for the pelvicfloor, thus promoting motivation and adherence to treatment. The hypothesis of this study is to prove that the use of a pelvicfloor medical device combined with 2 rehabilitation sessions is not inferior to pelvic-perineal rehabilitation.

DETAILED DESCRIPTION:
Two groups will be studied:

* the control group will undergo 15 sessions of pelvic-perineal rehabilitation, corresponding to the gold standard.
* the intervention group will use the medical device 3 times a week for 15 minutes over a 3-month period, in addition to 2 rehabilitation sessions. The participant will then be able to modify her program according to her symptoms.

Recruitment will be carried out with the help of healthcare professionals. The investigators involved in the study will be physiotherapists specializing in pelvic-perineal rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate, severe or very severe stress urinary incontinence or mixed stress urinary incontinence (according to ICIQ-UI SF questionnaire score: moderate (6-12), severe (13-18) and very severe (19-21))
* Patient aged between 18 and 60
* Patient with a quality of life score measured with the I-QoL questionnaire less than or equal to 70 (score measured from 0 to 100, with poor quality of life: 0-35; average quality of life: 36-70; good quality of life: 71-100)
* Not to have given birth in the last 6 months (to avoid post-partum physiological recovery)
* Signed informed consent
* Effective contraception throughout the study (declarative)
* Patient must have a smartphone running at least Android 7 and iOS 12
* Patient must be able to read and write French

Exclusion Criteria:

* Patients with mild stress urinary incontinence or mixed stress urinary incontinence (ICIQ-UI SF score: mild (1-5))
* Patient with a quality of life score above 70 (according to the I-QoL questionnaire: good quality of life: 71-100)
* Patient undergoing other pelvic-perineal rehabilitation during the study period
* Patients with neurological disease or congenital malformation, surgically or medically treated urinary incontinence or prolapse, perineal hypoesthesia or local conditions prohibiting the use of an intravaginal catheter
* Infection of the bladder or vagina, or any symptoms associated with infection (itching, pain on urination or fever)
* Contraindications to the use of the medical device
* Anatomy making catheter placement difficult or impossible; in the case of prolapse, specialist advice is recommended.
* Hemorrhage
* Patients with genitourinary cancer (within the last 5 years)
* Patients with extra-urethral "incontinence" (fistula, ectopic ureter)
* Patients with severe urinary retention
* Patient with vesico-ureteral reflux
* Patients with hypoactive bladder
* In case of peripheral denervation in the pelvic-perineal area, specialist advice is recommended
* Patients wearing a sacral neuromodulation device
* Patients in an exclusion period (determined by a previous or current study)
* Impossibility of giving the subject clear information (subject in an emergency situation, difficulties in understanding the subject, etc.)
* Patient under court protection
* Patient under guardianship or curatorship
* Pregnancy (positive pregnancy test)
* Breastfeeding (as the hormonal impregnation caused by breastfeeding has a negative impact on perineal tone)
* Use of Huawei and Oppo smartphones

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Urinary symptoms using the ICIQ-UI SF questionnaire | 6 months
  The non-inferiority of 2 sessions of pelvic floor rehabilitation associated with the use of the EMY medical device compared with 15 sessions of pelvic floor rehabilitation (gold standard) on the urinary symptoms score at 6 months will be assessed using the ICIQ-UI SF questionnaire.

SECONDARY OUTCOMES:
Quality of life using the I-QoL questionnaire | 0 month, 1 month, 3 months, 6 months, 12 months
  changes in quality of life will be studied using the validated I - QoL questionnaire
Urinary symptoms using the ICIQ-UI SF questionnaire | 0 month, 1 month, 3 months, 12 months
  changes in urinary symptoms will be studied using the validated ICIQ-UI SF questionnaire
Cost-utility ratio using the EQ-5D questionnaire | 0 month, 1 month, 3 months, 6 months, 12 months
  The cost/utility ratio will be studied using the cost/QALY ratio. The costs will relate to the consumption of reimbursed or non-reimbursed care (medical and paramedical consultations, hospitalization, drug treatment, absorbent pads, pessaries, etc.). QALYs will be estimated on the basis of responses to the validated EQ-5D 5L questionnaire.
Qualitative component | 1 month, 3 months, 6 months, 12 months
  the qualitative component will consist of questionnaires evaluating :
  * consumption of care at M0, M1, M3, M6 and M12 ;
  * ease of access to care at M1 ;
  * treatment satisfaction with the standardized PGI-I questionnaire and the question "do you recommend your treatment to a friend ?" at M3;
  * treatment adherence using a diary and a Likert scale between M0 and M3